CLINICAL TRIAL: NCT02504190
Title: Non-interventional Study Evaluating Efficacy and Tolerance on TEAM Conditioning (Thiotepa/Etoposide/Aracytin/Melphalan) Followed by Autologous Haematopoietic Stem Cells Transplantation in Patients With Lymphoma
Brief Title: Non-interventional Study on TEAM Conditioning in Patients With Lymphoma (TEAM)
Acronym: TEAM
Status: Completed | Type: Observational
Sponsor: Association for Training, Education, and Research in Hematology, Immunology, and Transplantation (Other)
Responsible Party: Sponsor
Other Study IDs: TEAM
Record Dates: First submitted 2015-07-20; First posted 2015-07-21 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Lymphoma
Keywords: Lymphoma; TEAM conditioning; autologous stem cells transplantation
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- lymphoma patients eligible for TEAM conditioning: Lymphoma Patients who are eligible will be included. Patients will undergo TEAM conditioning regimen followed by autologous haematopoietic stem cells transplantation according to standard practice of the centre and drugs label in France.

SUMMARY:
Lymphoma is a malignant blood disease sensitive to chemotherapy. In case of relapse after first-line treatment, high-dose chemotherapy conditioning followed by autologous hematopoietic stem cell transplantation (auto-HSCT) improves patient survival and reduces the risk of relapse. Auto-HSCT may also be indicated in the first line in case of aggressive lymphoma at high risk of relapse. BEAM (Carmustine, Etoposide, Aracytine and Melphalan) is the more frequently used high-dose conditioning regimen. Nevertheless, Carmustine is no longer available in Europe.

The investigators have therefore chosen to replace Carmustine by Thiotepa and use the TEAM regimen as the new conditioning. Indeed, Thiotepa is approved by french national agency for the security of drugs (ANSM) for use as part of auto-HSCT conditioning regimen. The results of TEAM regimen in terms of efficacy and toxicity appear similar to those of BEAM. However, no study have been performed prospectively. Only small series and case reports have been reported.

If the study confirms the results of retrospective studies, conditioning by TEAM could become a new standard in auto-HSCT for the treatment of lymphoma.

This study is non-interventional, prospective with 3 centers.

All included patients will receive, according to standard practice and drug label in France, the following diagram:

1. Conditioning:

   * Thiotepa 8 mg / kg to J-6
   * Etoposide 100 mg / m² / 12 h for 4 days (J-5 to D-2)
   * Aracytine 200 mg / m² / 12 h for 4 days (J-5 to D-2)
   * Melphalan 140 mg / m² on day-1
2. Transfusion graft: the day D0 with autologous peripheral stem cell transplant
3. Care supports: Patients will be treated according to the usual procedures of centers participating in the study at the discretion of the investigator.
4. Follow-up of patients will not be changed by the study.

The main objective of the study is to evaluate the progression-free survival (PFS) of lymphoma patients treated with autologous stem cells after conditioning by TEAM

Secondary objectives are:

* To evaluate overall survival;
* To assess the response to treatment;
* to evaluate the incidence of relapse;
* to assess the toxic transplant related mortality;
* to study transplant-related morbidity (infections, nutritional and gastrointestinal toxicity, immune reconstitution).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years,
* lymphoma confirmed by biopsy
* first autologous haematopoietic stem cells transplantation after TEAM conditioning

Exclusion Criteria:

* VIH, HBV, and/or HCV seropositive
* Contraindication to autologous stem cell transplantation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lymphoma patients will be recruited in on the French site
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2015-07-16 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 1 year after autologous haematopoietic stem cells transplantation

SECONDARY OUTCOMES:
Overall Survival | 100 days and at 1 year after autologous haematopoietic stem cells transplantation
Overall and complete response rate | 100 days and 1 year after autologous haematopoietic stem cells transplantation
Incidence of relapse | 100 days and 1 year after autologous haematopoietic stem cells transplantation
Impact of transplant-related mortality | 100 days and 1 year after autologous haematopoietic stem cells transplantation
Incidence of infections | during aplasia, 100 days and 1 year after autologous haematopoietic stem cells transplantation
Incidence of grade 3-4 side effects | during aplasia, 100 days and 1 year after autologous haematopoietic stem cells transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamad Mohty, Paris, France